CLINICAL TRIAL: NCT00583687
Title: Pulse Contour Analysis and Tissue Oxymetry in Changing Vascular Tone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Christoph C Ganter, MD, Departement of Intensive Care Medicine, University Hospital Inselspital, Berne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEK-3107-UHB-1316
Record Dates: First submitted 2007-12-18; First posted 2007-12-31 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Cardiac Output, High; Cardiac Output, Low; Vasodilation; Vasoconstriction; Hemodynamics
Keywords: Arterial pulse contour cardiac output; Changing vascular tone; Tissue Oxymetry; Prediction of Fluid Responsiveness
MeSH Terms: conditions — Cardiac Output, High; Cardiac Output, Low; Aneurysm | interventions — Spectroscopy, Near-Infrared

INTERVENTIONS:
Device: Vigileo TM / Flotrac TM (Minimally invasive cardiac output system consisting of arterial line sensor and cardiac output monitor) — Attachment of the arterial line sensor and pulse contour cardiac output monitor to the arterial line of the patient.
  Other Names: Vigileo TM / Flotrac TM
Other: Passive leg raising — Passive leg raising for prediction of fluid responsiveness with arterial pulse contour analysis.
Other: Volume challenge / Change of vasoactive drugs or inotropics — Either a volume challenge (using colloids or crystalloids) or a change in the dosage of of vasoactive drugs or inotropics, or a combination of them, as proposed by the treating physician.
Device: Inspectra TM/O-To-See TM (Tissue oxymetry with near infrared spectroscopy and laser-Doppler) — Tissue oxymetry continuously measured with near infrared spectrometry and laser Doppler during the whole study period.
  Other Names: Inspectra TM; O-To-See TM

SUMMARY:
The purpose of this study is to compare changes of minimally invasive arterial pulse contour cardiac output with changes of intermittent and continuous thermodilution cardiac output by pulmonary artery catheter in hemodynamic unstable patients with rapid changing vascular tone (changing dosage of vasoactive drugs or inotropics, or volume challenge). Simultaneously, global parameters of oxygen delivery and consumption will be compared with regional flow parameters and tissue oxymetry (near infrared spectrometry and laser-Doppler). While continuous thermodilution cardiac output is used for patient management, pulse contour cardiac output, intermittent thermodilution cardiac output and tissue oxymetry is only used for monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Indication for invasive hemodynamic monitoring with pulmonary artery catheter and arterial catheter
* Hemodynamic instability (need for vasoactive drugs, inotropics or volume).

Exclusion Criteria:

* Age < 18.
* Patient with contraindications for the placement of arterial cannula.
* Patient with history or clinical findings of aortic valve regurgitation.
* Atrial fibrillation.
* Patient being treated with an intra-aortic balloon pump.
* Limitation of therapy due to bad prognosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Changes of cardiac output measured by three different techniques during changes of vascular tone | 2 hours

SECONDARY OUTCOMES:
Prediction of fluid responsiveness with minimally invasive arterial pulse contour analysis in hemodynamic unstable patients. | 2 hours
Comparison of global parameters of oxygen delivery and consumption with local parameters of flow and tissue oxymetry during changes of vascular tone. | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christoph C Ganter, M.D., Principal Investigator — Department of Intensive Care Medicine, University Hospital, Inselspital, Berne
Locations (1):
- Department of Intensive Care Medicine, University Hospital Inselspital, Berne, Bern, Switzerland